CLINICAL TRIAL: NCT06507722
Title: Night Owl Metabolism: Investigating the Impact of Chronotype on Glucose Metabolism in Youth
Brief Title: Night Owl Metabolism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Lawson Wilkins Pediatric Endocrine Society (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); DexCom, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00428863
Record Dates: First submitted 2024-07-12; First posted 2024-07-18 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: PreDiabetes; Overweight; Impaired Glucose Tolerance
Keywords: chronotype; sleep
MeSH Terms: conditions — Prediabetic State; Overweight; Glucose Intolerance

STUDY DESIGN:
Intervention Model Description: For randomization in Aim 1, participants will be assigned to Early or Late OGTT for the first visit with crossover to the alternate for the second visit. In Aim 2, participants will be assigned to Early or Late standardized first meal for Day 1 with crossover to the alternate for Day 8.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Randomization will be done via a computer-generated random number list prepared by the statistician who will have no clinical involvement in the study. The list will then be provided to the study coordinator. The investigator will not be masked to assignment for Aim 1 as the investigator will be available during OGTT testing as needed. In Aim 2, the investigator will be blinded to randomization.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A - Late Chronotype first, then alternate (Other): Sleep onset after 2am
  Interventions: Diagnostic Test: Timing of OGTT; Behavioral: Timing of Standardized Meal
- Cohort B - Non-late Chronotype first, then alternate (Other): Sleep onset before 11pm
  Interventions: Diagnostic Test: Timing of OGTT; Behavioral: Timing of Standardized Meal

INTERVENTIONS:
Diagnostic Test: Timing of OGTT — In Aim 1, timing of oral glucose tolerance test will be altered.
Behavioral: Timing of Standardized Meal — In Aim 2, timing of a standardized meal will be altered.

SUMMARY:
The proposed study uses a novel and rigorous randomized cross-over study design in youth (17-23y) with late and non-late chronotype (n=35 per group) to assess the glycemic effect of "aligning" an oral glucose tolerance test (OGTT) or first-meal of day to a subject's chronotype. Both groups will undergo 2 OGTTs (aligned and mis-aligned with chronotype) to compare glucose tolerance and insulin sensitivity within-subject (primary outcome) and between groups (Aim 1). Then, youth will also undergo two standardized meals (aligned and mis-aligned with chronotype) while wearing continuous glucose monitoring to compare post-prandial glucose excursions within-subject and between groups (Aim 2). A pilot Exploratory Aim 3 (n=12 per group) will investigate delayed melatonin patterns under dim-light as a potential pathophysiologic mechanism behind abnormal glucose tolerance in youth with late chronotype on morning OGTTs.

ELIGIBILITY:
Inclusion Criteria:

* Overweight similar to (BMI ≥ 85th percentile but <95th percentile for age and sex per Centers for Disease Control and Prevention growth curves (as Centers for Disease Control and Prevention growth curves contain ages ≤ 20y; if ages 21-23 years, the BMI ≥ 85th and <95th percentile equivalents for a 20-year-old will be used))
* Post-pubertal
* Normal sleep duration (avg. >7 hours of sleep per night)
* Social jetlag (difference between weekend and weekday sleep) of < 2 hours.

Exclusion Criteria:

* Known diabetes, sleep disorders, major organ system illness, pregnancy, or genetic syndrome
* Medication use known to affect insulin sensitivity, glucose tolerance, or circadian rhythm
* Screening high risk for obstructive sleep apnea
* Night shift work.

Ages: 18 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
2-Hour Difference in Glucose | Day 4 and Day 11 of Aim 1 derived from OGTT
  Within-subject difference in 2-hour glucose after glucose ingestion on OGTT between early and late OGTT (primary analysis) in the late chronotype group and secondary analysis will be between group differences between early and late OGTT.
Insulin Sensitivity (by Oral Minimal Model) | Day 4 and Day 11 of Aim 1 derived from OGTT
  Within-subject difference in insulin sensitivity (derived from oral Minimal Model) between early and late OGTT (primary analysis) in the late chronotype group and secondary analysis will be between group differences between early and late OGTT.
2-hour Incremental Area Under the Curve (iAUC) for glucose | Day 1 and Day 8 of Aim 2 during post-prandial period following each standardized meal
  Within-subject difference in iAUC for glucose from continuous glucose monitor between early and late Meal (primary analysis) in the late chronotype group and secondary analysis will be between group differences between early and late Meal.

SECONDARY OUTCOMES:
Difference in Fasting Glucose | Day 4 and Day 11 of Aim 1 obtained before OGTT
  Within-subject difference in fasting glucose at start of OGTT between early and late OGTT (primary analysis) in the late chronotype group and secondary analysis will be between group differences between early and late OGTT.
Insulin secretion indices | Day 4 and Day 11 of Aim 1 derived from OGTT
  Within-subject difference in insulin secretion (dynamic phase, static phase, total and insulin secretory rate) from c-peptide minimal model between early and late OGTT (primary analysis) in the late chronotype group and secondary analysis will be between group differences between early and late OGTT.
Incremental Area Under the Curve (iAUC) for Insulin | Day 4 and Day 11 of Aim 1 derived from OGTT
  Within-subject difference in iAUC for insulin after glucose ingestion between early and late OGTT (primary analysis) in the late chronotype group and secondary analysis will be between group differences between early and late OGTT.
Hemoglobin A1c levels | Day 4 of Aim 1 during first OGTT Visit
  Analysis of between group differences in hemoglobin A1c levels
Difference in Disposition Index | Day 4 and Day 11 of Aim 1 derived from OGTT
  Within-subject difference in disposition index (derived from insulin sensitivity and insulin secretion metrics) between early and late OGTT (primary analysis) in the late chronotype group and secondary analysis will be between group differences between early and late OGTT.
Difference in Insulin Clearance | Day 4 and Day 11 of Aim 1 derived from OGTT
  Within-subject difference in insulin clearance (derived from Watanabe et al. model) between early and late OGTT (primary analysis) in the late chronotype group and secondary analysis will be between group differences between early and late OGTT.
Mean Glucose | Up to 8 days
  Analysis of between group differences in mean glucose derived from continuous glucose monitor
Percent Time Spent Above 120 mg/dL | Up to 8 days
  Analysis of between group differences in time spent above 120 mg/dL derived from continuous glucose monitor. Over course of wearing continuous glucose monitor for Aim 2 (8 days)]
Percent Time Spent Above 140 mg/dL | Up to 8 days
  Analysis of between group differences in time spent above 140 mg/dL derived from continuous glucose monitor. Over course of wearing continuous glucose monitor for Aim 2 (8 days).
Number of Excursions greater than 140mg/dL | Up to 8 days
  Analysis of between group differences in the number of excursions above 140 mg/dL derived from continuous glucose monitor. Over course of wearing continuous glucose monitor for Aim 2 (8 days).
Difference in Post-prandial peak | Day 1 and Day 8 of Aim 2 during post-prandial period following each standardized meal
  Within-subject difference in post-prandial peak from continuous glucose monitor between early and late Meal (primary analysis) in the late chronotype group and secondary analysis will be between group differences between early and late Meal
Standard Deviation of Glucose | Up to 8 days
  Analysis of between group differences in standard deviation of glucose derived from continuous glucose monitor. Over course of wearing continuous glucose monitor for Aim 2 (8 days).
Coefficient of Variation of Glucose | Up to 8 days
  Analysis of between group differences in coefficient of variation of glucose derived from continuous glucose monitor. Over course of wearing continuous glucose monitor for Aim 2 (8 days).

CONTACTS AND LOCATIONS:
Overall Officials: Talia Hitt, MD/MPH/MSHP, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins School of Medicine, Baltimore, Maryland, United States

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-01-30): https://cdn.clinicaltrials.gov/large-docs/22/NCT06507722/Prot_SAP_001.pdf
  • Informed Consent Form (2024-10-15): https://cdn.clinicaltrials.gov/large-docs/22/NCT06507722/ICF_002.pdf